CLINICAL TRIAL: NCT04608994
Title: Long-term Follow-up in Survivors of Critical Illness: An Longitudinal Assessment of Critically Ill Patients Discharged Alive From the Intensive Care Unit
Brief Title: Long-term Follow up in Survivors of Critical Illness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Piva Simone, Principal Investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: NP2595
Record Dates: First submitted 2020-10-03; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Post Intensive Care Unit Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Survivors of critical illness may suffer from persistent physical, cognitive and mental impairments, such as muscle weakness, dysfunction in the memory and executive domains, post-traumatic stress disorders, depression, and anxiety. This syndrome is referred to as Post Intensive Care Syndrome (PICS).

This study aims to assess the frequency of impairments, their evolution over time, and to understand the pathogenetic mechanisms and the association between long-term sequelae and acute care events.

DETAILED DESCRIPTION:
PICS describes 'new or worsening impairments in physical, cognitive or mental health status arising after critical illness and persisting beyond acute care hospitalization'. Different critical care professional and scientific societies have identified long-term functional outcomes after critical illness as an important target for research and clinical improvements, and there is general agreement that research on PICS should be a priority for the critical care community.

Post-ICU subjects may experience physical problems, such as muscles weakness and wasting, caused by prolonged bed rest and immobility during the ICU stay and by critical illness polyneuropathy and myopathy developing during the acute illness; organ dysfunction; chronic pain; mental health problems including depression, anxiety or post-traumatic stress disorder (PTSD); and neurocognitive impairments which are predominantly represented by memory dysfunction and executive function impairment. The impact of these problems on the subject's health status is huge, which reduced quality of life, and impaired functional status, and daily functioning.

Many survivors incur substantial healthcare costs, lose employment, and find their social networks wholly changed. The costs to subjects and families are high: ICU survivorship is associated with decreased return to work, and the loss of earnings plagues both patients and caregivers.

Prior studies in which researchers have examined outcomes among ICU survivors have been mainly restricted their assessments to specific patient populations and have used only limited outcome measures or the follow-up period was relatively short-term. Moreover, few studies have explored the association between acute care events and long-term sequelae as well as the underlying pathophysiological mechanisms.

The researchers appertaining to the present study implemented a follow-up clinic to describe the frequency of physical, cognitive, and mental impairments and their evolution over time in subjects surviving critical illness. The researchers also aim at understanding the pathogenetic mechanisms underlying these impairments and their association with acute care events.

ELIGIBILITY:
Inclusion Criteria:

- All COVID-19 patients admitted to the ICUs of the Spedali Civili University Hospital in Brescia, Italy.

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will enroll all patients admitted to the ICUs with SARS-CoV-2 pneumonia and ARDS.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Medical Research Council (MRC) sum score | 3 months
  Medical Research Council (MRC)-sum score evaluates global muscle strength, and it has been proposed in PICS syndrome post-COVID-19. Manual strength of six muscle groups (shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and ankle dorsiflexion) is evaluated on both sides using the MRC-sumscore. The summation of scores gives MRC-sumscore, ranging from 0 to 60. This score reliably identifies significant weakness (< 48) and even better in severe weakness (<36).
Medical Research Council (MRC) sum score | 6 months
  Medical Research Council (MRC)-sum score evaluates global muscle strength, and it has been proposed in PICS syndrome post-COVID-19. Manual strength of six muscle groups (shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and ankle dorsiflexion) is evaluated on both sides using the MRC-sumscore. The summation of scores gives MRC-sumscore, ranging from 0 to 60. This score reliably identifies significant weakness (< 48) and even better in severe weakness (<36).
Medical Research Council (MRC) sum score | 12 months
  Medical Research Council (MRC)-sum score evaluates global muscle strength, and it has been proposed in PICS syndrome post-COVID-19. Manual strength of six muscle groups (shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and ankle dorsiflexion) is evaluated on both sides using the MRC-sumscore. The summation of scores gives MRC-sumscore, ranging from 0 to 60. This score reliably identifies significant weakness (< 48) and even better in severe weakness (<36).
Dominand Handgrip Test | 3 months
  Dynamometry will be considered normal if >11Kg in Male and 7.5 kg in Female. Moreover, the researcher will standardized the result as percentage of the predicted normal value (PNV) as follow: <20% PNV; 20%<=PNV< 40%; 40%<=PNV< 60%; 60%<= PNV< 80%, and >=80 PNV. [DOI: 10.1016/j.clnu.2008.04.004]
Dominand Handgrip Test | 6 months
  Dynamometry will be considered normal if >11Kg in Male and 7.5 kg in Female. Moreover, the researcher will standardized the result as percentage of the predicted normal value (PNV) as follow: <20% PNV; 20%<=PNV< 40%; 40%<=PNV< 60%; 60%<= PNV< 80%, and >=80 PNV. [DOI: 10.1016/j.clnu.2008.04.004]
Dominand Handgrip Test | 12 months
  Dynamometry will be considered normal if >11Kg in Male and 7.5 kg in Female. Moreover, the researcher will standardized the result as percentage of the predicted normal value (PNV) as follow: <20% PNV; 20%<=PNV< 40%; 40%<=PNV< 60%; 60%<= PNV< 80%, and >=80 PNV. [DOI: 10.1016/j.clnu.2008.04.004]
Six Minutes Walking Test | 3 months
  Six-minute walking test will be performed in accordance with the America Thoracic Society recommendations and it will be adjusted for age, sex, height, and body weight
Six Minutes Walking Test | 6 months
  Six-minute walking test will be performed in accordance with the America Thoracic Society recommendations and it will be adjusted for age, sex, height, and body weight
SIX Minutes Walking Test | 12 months
  Six-minute walking test will be performed in accordance with the America Thoracic Society recommendations and it will be adjusted for age, sex, height, and body weight
Fatigue Severity Scale (FSS) | 3 months
  The Fatigue severity score is a nine-item unidimensional questionnaire that measures the severity of fatigue symptoms on a seven-point ordinal scale (maximum score of seven). An FSS ≥36 will be considered as an indicator of fatigue.
Fatigue Severity Scale (FSS) | 6 months
  The Fatigue severity score is a nine-item unidimensional questionnaire that measures the severity of fatigue symptoms on a seven-point ordinal scale (maximum score of seven). An FSS ≥36 will be considered as an indicator of fatigue.
Fatigue Severity Scale (FSS) | 12 months
  The Fatigue severity score is a nine-item unidimensional questionnaire that measures the severity of fatigue symptoms on a seven-point ordinal scale (maximum score of seven). An FSS ≥36 will be considered as an indicator of fatigue.
Elettromyography | 3 months
  Simplified peroneal nerve test (PENT)wiil be used to diagnose a critical illness polyneuropathy and myopathy; a value <5.26 mV present in both legs was considered as abnormal.
Elettromyography | 6 months
  Simplified peroneal nerve test (PENT)wiil be used to diagnose a critical illness polyneuropathy and myopathy; a value <5.26 mV present in both legs was considered as abnormal.
Elettromyography | 12 months
  Simplified peroneal nerve test (PENT)wiil be used to diagnose a critical illness polyneuropathy and myopathy; a value <5.26 mV present in both legs was considered as abnormal.
Montreal Cognitive Assessment Test (MoCA) | 3 months
  Montreal Cognitive Assessment (MoCA) is divided into several cognitive domains with variable scoring among them, adding up to a maximum total of 30 points if all responses are correct. The scale is divided into Visuospatial and executive functioning (5 points), animal naming (3 points), attention (6 points), language (3 points), abstraction (2 points), delayed recall (short-term memory, 5 points), and orientation (6 points). To correct for educational effects found in the original study, one point is added if the subject has less than 12 years of education. The suggested cutoff score for normalcy in the MoCA is 26/30. When patients scored less than 26, we used the following classification: 18-25 = mild cognitive impairment, 10-17= moderate cognitive impairment, and less than 10= severe cognitive impairment
Montreal Cognitive Assessment Test (MoCA) | 6 months
  Montreal Cognitive Assessment (MoCA) is divided into several cognitive domains with variable scoring among them, adding up to a maximum total of 30 points if all responses are correct. The scale is divided into Visuospatial and executive functioning (5 points), animal naming (3 points), attention (6 points), language (3 points), abstraction (2 points), delayed recall (short-term memory, 5 points), and orientation (6 points). To correct for educational effects found in the original study, one point is added if the subject has less than 12 years of education. The suggested cutoff score for normalcy in the MoCA is 26/30. When patients scored less than 26, we used the following classification: 18-25 = mild cognitive impairment, 10-17= moderate cognitive impairment, and less than 10= severe cognitive impairment
Montreal Cognitive Assessment Test (MoCA) | 12 months
  Montreal Cognitive Assessment (MoCA) is divided into several cognitive domains with variable scoring among them, adding up to a maximum total of 30 points if all responses are correct. The scale is divided into Visuospatial and executive functioning (5 points), animal naming (3 points), attention (6 points), language (3 points), abstraction (2 points), delayed recall (short-term memory, 5 points), and orientation (6 points). To correct for educational effects found in the original study, one point is added if the subject has less than 12 years of education. The suggested cutoff score for normalcy in the MoCA is 26/30. When patients scored less than 26, we used the following classification: 18-25 = mild cognitive impairment, 10-17= moderate cognitive impairment, and less than 10= severe cognitive impairment
Hospital Anxiety and Depression Scale (HADS) | 3 months
  Hospital Anxiety and Depression Scale (HADS) was classified as follow: HADS for depression: 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case) and HADS Anxiety: 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case).
Hospital Anxiety and Depression Scale (HADS) | 6 months
  Hospital Anxiety and Depression Scale (HADS) was classified as follow: HADS for depression: 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case) and HADS Anxiety: 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case).
Hospital Anxiety and Depression Scale (HADS) | 12 months
  Hospital Anxiety and Depression Scale (HADS) was classified as follow: HADS for depression: 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case) and HADS Anxiety: 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case).
The The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | 3 months
  The PCL-5 is a self-report measure that assesses the presence and severity of Post Traumatic Stress Disorder (PTSD) symptoms. Items on the PCL-5 correspond with DSM-5 criteria for PTSD. PTSD >32 is strongly associated with the presence of PTSD.
The The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | 6 months
  The PCL-5 is a self-report measure that assesses the presence and severity of Post Traumatic Stress Disorder (PTSD) symptoms. Items on the PCL-5 correspond with DSM-5 criteria for PTSD. PTSD >32 is strongly associated with the presence of PTSD.
The The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | 12 months
  The PCL-5 is a self-report measure that assesses the presence and severity of Post Traumatic Stress Disorder (PTSD) symptoms. Items on the PCL-5 correspond with DSM-5 criteria for PTSD. PTSD >32 is strongly associated with the presence of PTSD.
Insomnia Severity Index (ISI) | 3 months
  Insomnia Severity Index (ISI) is a brief instrument that was designed to assess the severity of both nighttime and daytime components of insomnia. It is available in several languages and is increasingly used as a metric of treatment response in clinical research. ISI will be classified as follows: No clinically significant insomnia (0-7), Subthreshold insomnia (8-14), Moderate insomnia (15-21), and severe insomnia (22-28).
Insomnia Severity Index (ISI) | 6 months
  Insomnia Severity Index (ISI) is a brief instrument that was designed to assess the severity of both nighttime and daytime components of insomnia. It is available in several languages and is increasingly used as a metric of treatment response in clinical research. ISI will be classified as follows: No clinically significant insomnia (0-7), Subthreshold insomnia (8-14), Moderate insomnia (15-21), and severe insomnia (22-28).
Insomnia Severity Index (ISI) | 12 months
  Insomnia Severity Index (ISI) is a brief instrument that was designed to assess the severity of both nighttime and daytime components of insomnia. It is available in several languages and is increasingly used as a metric of treatment response in clinical research. ISI will be classified as follows: No clinically significant insomnia (0-7), Subthreshold insomnia (8-14), Moderate insomnia (15-21), and severe insomnia (22-28).
The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) | 3 months
  The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) is a widely used and extensively validated generic QOL measure that consists of 8 multiple-item domains. We applied two different methods for scoring. Firstly, for each item, a scale between 0-100 will be calculated and the percentage of predicted value has been calculated, based on the Italian normalized value.
  The second method will be been the calculation ofthe physical component summary (PCS) and the mental component summary (MCS), as described by Taft et al. After the eight scale scores are calculated, a z-score is determined for each by subtracting the scale mean of a sample of the Italian general population from an individual's scale score and then dividing by the standard deviation from the Italian general population. Each of the eight z-scores is then multiplied by the corresponding factor scoring coefficient for the scale.
The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) | 6 months
  The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) is a widely used and extensively validated generic QOL measure that consists of 8 multiple-item domains. We applied two different methods for scoring. Firstly, for each item, a scale between 0-100 will be calculated and the percentage of predicted value has been calculated, based on the Italian normalized value.
  The second method will be been the calculation ofthe physical component summary (PCS) and the mental component summary (MCS), as described by Taft et al. After the eight scale scores are calculated, a z-score is determined for each by subtracting the scale mean of a sample of the Italian general population from an individual's scale score and then dividing by the standard deviation from the Italian general population. Each of the eight z-scores is then multiplied by the corresponding factor scoring coefficient for the scale.
The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) | 12 months
  The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) is a widely used and extensively validated generic QOL measure that consists of 8 multiple-item domains. We applied two different methods for scoring. Firstly, for each item, a scale between 0-100 will be calculated and the percentage of predicted value has been calculated, based on the Italian normalized value.
  The second method will be been the calculation ofthe physical component summary (PCS) and the mental component summary (MCS), as described by Taft et al. After the eight scale scores are calculated, a z-score is determined for each by subtracting the scale mean of a sample of the Italian general population from an individual's scale score and then dividing by the standard deviation from the Italian general population. Each of the eight z-scores is then multiplied by the corresponding factor scoring coefficient for the scale.
Barthel Index (BI) | 3 months
  BI will be classified as follow: Independent (80-100); Minimally dependent (60-79);, Partially dependent (40-59), Very dependent (20-39); and Totally dependent (<20).
Barthel Index (BI) | 6 months
  BI will be classified as follow: Independent (80-100); Minimally dependent (60-79);, Partially dependent (40-59), Very dependent (20-39); and Totally dependent (<20).
Barthel Index (BI) | 12 months
  BI will be classified as follow: Independent (80-100); Minimally dependent (60-79);, Partially dependent (40-59), Very dependent (20-39); and Totally dependent (<20).

CONTACTS AND LOCATIONS:
Locations (1):
- ASST- Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Derived] Latronico N, Peli E, Calza S, Rodella F, Novelli MP, Cella A, Marshall J, Needham DM, Rasulo FA, Piva S; LOTO Investigators. Physical, cognitive and mental health outcomes in 1-year survivors of COVID-19-associated ARDS. Thorax. 2022 Mar;77(3):300-303. doi: 10.1136/thoraxjnl-2021-218064. Epub 2021 Sep 29. PMID 34588274